CLINICAL TRIAL: NCT01185392
Title: European Cardiac Resynchronisation Therapy Survey
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Boston Scientific Corporation (Industry); Medtronic (Industry); Abbott Medical Devices (Industry); Biotronik SE & Co. KG (Industry); LivaNova (Industry); Roche Diagnostic Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CRT Survey
Record Dates: First submitted 2010-08-07; First posted 2010-08-19 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2012-06

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronisation Therapy in Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The European CRT survey represents a joint initiative between two ESC associations; the Heart Failure Association and the European Heart Rhythm Association. The survey will be performed in collaboration with The Institute für Herzinfarktforschung in Ludwigshafen which will handle the data collection and data analysis.

DETAILED DESCRIPTION:
This European CRT Survey was initiated by the Heart Failure Association (HFA) and the European Heart Rhythm Association (EHRA) of the ESC in order to describe current European practice and routines associated with CRT-P/CRT-D implantations based on sample of patients enrolled in 13 countries. The data collected following implantation provides information including clinical characteristics, diagnostic criteria, implantation routines and techniques, adverse experience, and assessment of adherence to guideline recommendations. The single follow-up visit at 1 year (9-15 months) will provide information regarding short-term clinical outcomes.

The primary objective of this Survey is to describe current European practice based on a broad sampling in 13 countries. The information collected will enable practice between centres and countries to be compared and permit benchmarking with national and international practice. The survey provides valuable quality assurance assessment for individual centres, permits limited economic analyses and broadly evaluates adherence to guideline recommendations.

The following 13 European countries contributed patients to the survey: Austria, Belgium, France, Germany, Ireland, Israel, Italy, the Netherlands, Norway, Spain, Sweden, Switzerland and UK. Two national coordinators, one each from the fields of heart failure and electrophysiology, were selected and given the responsibility to facilitate recruitment in their respective countries.

Follow the link for complete list of the members of the Scientific Committee and national coordinators.

ELIGIBILITY:
Inclusion Criteria:

* eligible patients for CRT-P or CRT-D.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients successfully implanted with a new CRT-P, CRT-D or upgrades during the inclusion period were eligible. The successful procedure itself identified the patient as a survey candidate. Patients screened but not successfully implanted were not entered into the survey. Ethics approval and written informed consent were obtained in countries where required.
Sampling Method: Non-Probability Sample
Enrollment: 2438 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To describe current European CRT implantation practice and there is a need to precisely quantify the extent of treatment failures, adverse experience and complications associated with implantation. | November 2008-October 2010
  The Survey will capture data from patients receiving CRT-P/CRT-D devises:
  * Demographics and clinical characteristics
  * Diagnostic criteria assessed prior to implantation
  * Pharmacological therapy at baseline and follow-up
  * Implantation procedure and techniques
  * Device programming
  * Short and long-term outcomes
  * Adverse experience and hospitalisation
  * Economic analyses
  * Adherence to guidelines
  These data should also provide information contrasting practice between centres and countries and adherence to guideline recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Dickstein, MD, PHD, Study Chair — HFA of the ESC; Silvia Priori, MD, PHD, Study Chair — EHRA of the ESC; Angelo Auricchio, MD, PHD, Study Director — EHRA of the ESC; Josep Brugada, MD, PHD, Study Director — EHRA of the ESC; John Cleland, MD, PHD, Study Director — HFA of the ESC; Geneviève Derumeaux, MD, PHD, Study Director — EAE of the ESC; Daniel Gras, MD, PHD, Study Director — EHRA of the ESC; Michel Komajda, MD, PHD, Study Director — HFA of the ESC; Cecilia Linde, MD, PHD, Study Director — EHRA of the ESC; John Morgan, MD, PHD, Study Director — EHRA of the ESC; Dirk J van Veldhuisen, MD, PHD, Study Director — HFA of the ESC; Anselm Gitt, MD, Study Director — The Institut für Herzinfarktforschung in Ludwigshafen, Germany; Nigussie Bogale, MD, Study Director — Stavanger University Hospital and University of Bergen, Norway

REFERENCES:
- [Background] CRT Survey Scientific Committee. European cardiac resynchronization therapy survey: rationale and design. Eur J Heart Fail. 2009 Mar;11(3):326-30. doi: 10.1093/eurjhf/hfp030. PMID 19228801
- [Result] Dickstein K, Bogale N, Priori S, Auricchio A, Cleland JG, Gitt A, Limbourg T, Linde C, van Veldhuisen DJ, Brugada J; Scientific Committee; National Coordinators. The European cardiac resynchronization therapy survey. Eur Heart J. 2009 Oct;30(20):2450-60. doi: 10.1093/eurheartj/ehp359. Epub 2009 Aug 31. PMID 19723694
- [Derived] Bogale N, Priori S, Cleland JG, Brugada J, Linde C, Auricchio A, van Veldhuisen DJ, Limbourg T, Gitt A, Gras D, Stellbrink C, Gasparini M, Metra M, Derumeaux G, Gadler F, Buga L, Dickstein K; Scientific Committee, National Coordinators, and Investigators. The European CRT Survey: 1 year (9-15 months) follow-up results. Eur J Heart Fail. 2012 Jan;14(1):61-73. doi: 10.1093/eurjhf/hfr158. PMID 22179034
- [Derived] Bogale N, Witte K, Priori S, Cleland J, Auricchio A, Gadler F, Gitt A, Limbourg T, Linde C, Dickstein K; Scientific Committee, National coordinators and the investigators. The European Cardiac Resynchronization Therapy Survey: comparison of outcomes between de novo cardiac resynchronization therapy implantations and upgrades. Eur J Heart Fail. 2011 Sep;13(9):974-83. doi: 10.1093/eurjhf/hfr085. Epub 2011 Jul 19. PMID 21771823
- See also: Synopsis of the Survey, list of participating countries and members of the Scientific Committee and national coordinators — http://www.crt-survey.org